CLINICAL TRIAL: NCT05574465
Title: Esophageal Manometry During Recovery From Endotracheal Intubation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-36634
Record Dates: First submitted 2022-04-21; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Motility Function
Keywords: Extubation; Manometry

STUDY DESIGN:
Intervention Model Description: Subjects who meet the inclusion and exclusion criteria will be eligible for participation in this study. It is anticipated that the largest number of subjects will come from patients undergoing extubation in an intensive care unit (ICU).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Manometry Device (Other): At 10 minutes prior to anticipated removal of the endotracheal tube, pass the routine manometry catheter per naris to 30 cms.
  Interventions: Device: High resolution solid state manometry

INTERVENTIONS:
Device: High resolution solid state manometry — The use of esophageal manometry device during removal of endotracheal tube by anesthesia

SUMMARY:
1. An intact pharyngoesophageal reflex is essential to protect the upper airway from aspiration of either mouth contents or regurgitated gastric refluxate. This reflex is essential at protecting the airway in all patients.
2. In patients, while under medication to tolerate endotracheal intubation, it is postulated that an identifiable upper esophageal sphincter and esophageal peristalsis are not present.
3. With the cessation of anesthetics, accompanied by the reversal of nerve block, normal pharyngoesophageal peristaltic activity correlates with awakening the patient from anesthesia. This would be identified by the performance of esophageal manometry.
4. A return of normal verbally stimulated pharyngoesophageal swallowing sequence accurately identifies a safe time to remove endotracheal tubes and/or reverse anesthesia. This verbally stimulated swallowing sequence correlated precisely with the return of objective pharyngoesophageal function.

DETAILED DESCRIPTION:
The emergence from routine general deep anesthesia with an endotracheal tube is a potentially dangerous time for patients. Patients cannot reliably maintain competence of the upper esophageal sphincter, thus aspiration of the contents from the mouth or regurgitated material from the stomach can be aspirated into the lungs leading to serious complications. In normal awake individuals the upper esophageal sphincter (also known as the cricopharyngeus or the inferior pharyngeal constrictor) is contracted and relaxes precisely timed with voluntary or involuntary swallowing. The swallowing sequence in normal awake persons begins with 1) the contraction of the upper and middle pharyngeal constrictors, 2) the posterior movement of the tongue and 3) the prompt relaxation of the contracted upper esophageal sphincter. Peristalsis then begins in the body of the esophagus leading contents to the stomach. The above is the normal sequence in humans, a process which maintains absolute separation of the airway and digestive passageways despite being in intimate proximity. During the early period of emergence from anesthesia, the aspiration risk is highest due to the sluggish return of the resting pressure in the upper esophagus and the lack of normal coordination with involuntary swallowing. Thus patients can't protect their airway by maintaining competence and appropriate relaxation of the upper esophageal sphincter. Routine high resolution solid state manometry is a standard routine technique is currently performed in awake patients sitting upright voluntarily requested to swallow small boluses of liquid. The entire sequence of events is studied using high resolution solid state manometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age (ASA I or II).
* Already scheduled for endotracheal tube extubation.
* Willing and able to give informed consent in either English or Spanish.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Patients not meeting entry criteria above.
* Refusal to give informed consent.
* Coagulopathy (INR > 2 and/or platelet count < 100,000.
* White Blood Cell count < 5,000/mm3
* Arrhythmia
* Serum creatinine > 2 mg/dl
* Prior known or suspected nasal obstruction.
* Known or suspected Zenker's diverticulum of esophagus, esophageal stricture, head/neck radiation therapy, hereditary telangiectasis, esophageal varices, cirrhosis.
* Anticoagulant usage such as heparin or Plavix

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The Basal Pressures of patients during High-Resolution Motility/Manometry (HRM): | The change in Basal Pressures will be recorded at the end of procedure.
  High-resolution manometry (HRM) determination of return of cricopharyngeal function
  - Basal Pressures: Upper esophageal sphincter (mmHg) - normal (34-104)
The Residual Pressures of patients during High-Resolution Motility/Manometry (HRM): | The change in Residual Pressures will be recorded at the end of procedure.
  - Residual Pressures: Upper esophageal sphincter (mmHg) - normal (<12.0)
The Wave Duration of patients during High-Resolution Motility/Manometry (HRM): | The change in Wave Duration will be recorded at the end of procedure.
  - Motility: Wave Duration (seconds) - normal (2.7-5.4)

SECONDARY OUTCOMES:
Percentage of patients agreeing to study versus refusing study. | During enrollment
  Percentage/number of patients/next of kin accepting protocol
Number of patients completing study. | At the completion of procedure
  Percentage/number of patients completing esophageal motility/manometry study.
Duration of HRM | The HRM study of the cricopharyngeus will be measured for the 5 minute time period just before planned endotracheal extubation to the time during extubation and for the 5 minute period just after endotracheal extubation.
  Duration (minutes) of motility/manometry research study during withdrawal of endotracheal intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Rogers, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No